CLINICAL TRIAL: NCT04827225
Title: Assessment of the Mental State of Parents of Premature Children and Impact on Neurodevelopment of the Child (Parents Psychic Preterm)
Brief Title: Assessment of the Mental State of Parents of Premature Children and Impact on Neurodevelopment of the Child
Acronym: PoPPY
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC20_0132
Record Dates: First submitted 2020-09-01; First posted 2021-04-01 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Parent-Child Relations
Keywords: prematurity; psychic state
MeSH Terms: conditions — Premature Birth | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PoPPY Group: Mother, Father and child born prematurely
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — Questionnaires (EPDS, HADS, PPQ, MIBS, etc.) will have to be completed by the parents at different stages of their child's development (38 weeks of amenorrhea, 3 months and 24 months).

SUMMARY:
The objective of the study is to assess the psychic profile of parents of children born prematurely

DETAILED DESCRIPTION:
Prematurity affects aroound 1 in 10 children worlwide. Many studies have shown the role of prematurity in the development of depression, anxiety, post-traumatic stress disorder, mother-to-child attachment disorders, but few studies have sought to assess the evolution of this profile over time as well as to assess all of the parents' psychic dimensions.

The investigators currently have little knowledge of risk factors (psychological or psychiatric history, follow-up undertaken, treatments implemented, etc.) that may favor the occurrence of postpartum mental disorders (anxiety, depression, post-traumatic stress disorder ).

The investigators will thus seek to identify them. Prematurity can have a negative impact on the parents' psychic experience in the postpartum period. However, few studies have examined the evolution over time of the parental psychic profile and its possible repercussions on the child in terms of attachment and becoming neurodevelopmental. Finally, the majority of studies dealing with these subjects concern only mothers.Tthe investigators will endeavor here to also take into account the fathers.

ELIGIBILITY:
Inclusion Criteria:

Parents whose child meets the following criteria:

* Singleton child
* Child aged up to 40 weeks of amenorrhea of age corrected at the time of inclusion
* Premature child as defined below:

  * Born at a term less than or equal to 34 weeks of amenorrhea And or
  * weighing 1500g or less at birth
* Hospitalized in the neonatology department of the Angers University Hospital
* Child included in Réseau Grandir Ensemble (RGE) in Pays de la Loire
* Informed consent form signed by both parents for their participation and the collection of data from the RGE for the child

Non-inclusion Criteria:

* Parents not fluent in the French language, implying not being able to complete the various questionnaires
* Parents including the child :

  * Is from a twin pregnancy or more
  * Has polymalformative syndrome or chromosomal abnormalities

Exclusion Criteria:

- Death of the child or one of the parents during follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children born prematurely hospitalizes in the neonatalogy department of the Angers University Hospital and included in the cohort 'Réseau Grandir Ensemble en Pays de la Loire'.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Assessing the psychic profile of parents of children born prematurely | At 38 weeks of amenorrhea (+/- 2 weeks)
  The psychic profile of the parents will be evaluated from the score obtained in the following autoquestionnaire :
  - parental depression (Edinburgh Postnatal Depression Scale (EPDS)), a score greater than or equal to 10 is in favour of parental depression
Assessing the psychic profile of parents of children born prematurely | At 38 weeks of amenorrhea (+/- 2 weeks)
  The psychic profile of the parents will be evaluated from the score obtained in the following autoquestionnaire :
  - parental anxiety (Hospital Anxiety and Depression Scale (HADS)), a score greater than or equal to 11 of the sub-scale anxiety is in favor of a parental anxiety
Assessing the psychic profile of parents of children born prematurely | At 38 weeks of amenorrhea (+/- 2 weeks)
  The psychic profile of the parents will be evaluated from the score obtained in the following autoquestionnaire :
  - posttraumatic stress parental ( Perinatal Posttraumatic Stress disorder Questionnaire (PPQ)), a score greater than or equal to 6 is in favour of posttraumatic parental stress

SECONDARY OUTCOMES:
Study the evolution of parents' psychic profile over time | At 3 months corrected age and at 24 months corrected age
  Use of the same tools and criteria as at 38 weeks of amenorrhea (parental depression : score EPDS ≥ 10)
Study the evolution of parents' psychic profile over time | At 3 months corrected age and at 24 months corrected age
  Use of the same tools and criteria as at 38 weeks of amenorrhea (parental anxiety HADS ≥11)
Study the evolution of parents' psychic profile over time | At 3 months corrected age and at 24 months corrected age
  Use of the same tools and criteria as at 38 WA (posttraumatic stress parental : PPQ ≥ 6)
Investigate the presence of peritraumatic dissociation experiments | At 38 weeks of amenorrhea (+/- 2 weeks)
  A score greater than 15 from the PDEQ (Peritraumatic Dissociative Experiences Questionnaire) is considered a score in favour of a significant traumatic dissociation. Minimum scale value : 10, full scale value : 50. Abnormal if greater than or equal to 15.
Assess the mother's attachment to her child | At 38 weeks of amenorrhea and 3 months corrected age of the child
  A score equal to or greater than 2 from the MIBS questionnaire (Mother To Infant Bonding Scale) highlights mother-child disorders. This questionnaire is given only to the mother. Minimum scale value : 0, full scale value : 24. Abnormal if greater than or equal to 2.
Assess the parental stress | At 24 months corrected age
  A PSI (Parenting Stress Index) high score (percentile rank greater than or equal to 85) is considered a score in favour af a parental stress. Minimum scale value : 0, full scale value : 180. Abnormal if greater than or equal to 85.
study perinatal or prenatal psychological and psychiatric factors associated with depression, anxiety and post traumatic stress | at 38 weeks of amenorrhea (+/- 2 weeks), and 3 months corrected age and at 24 months corrected age
  these factors are studied by assessing whether or not there is a psychological and / or psychiatric history, medical-psychological follow-up, treatments taken.
Study the impact of the parental psychic profile on the neurological development of the child | At 24 months corrected age
  A ASQ (Ages Stages Questionnaire) score less than 185 is considered not optimal.
  The other data collected during the evaluation of the 24 months of age corrected as part of the Réseau Grandir Ensemble (RGE) will be used for the evaluation of neurological development. These data make it possible to classify children's development into optimal or non-optimal according to a rating system which has been defined by the network's scientific council.The impact of the parental psychic profile (at 38 WA +/- 2 weeks, at 3 months and at 24 months of their child's corrected age) on neurological development will be evaluated by Odds Ratios (ORs): ORs measuring the association between the parental psychic profile and the non-optimal ASQ score, ORs measuring the association between the parental psychic profile and the non-optimal development category according to the RGE rating.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France